CLINICAL TRIAL: NCT04801979
Title: Normative Values and Reference Equations of a New Incremental Step Test for the Assessment of Exercise Capacity for Portuguese Adults
Status: Completed | Type: Observational
Sponsor: Polytechnic Institute of Porto (Other)
Collaborators: Nippon Gases Portugal (Unknown)
Responsible Party: Principal Investigator, Rui Vilarinho, Principal Investigator, Polytechnic Institute of Porto
Other Study IDs: New_Step_Test
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Adults Without Disabilities
Keywords: Normative values; Reference equations; Step test; Exercise capacity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Incremental Step Test — Performance of the incremental step test (number of steps) for the assessment of exercise capacity. The step test will be designed according to the characteristics of other validated field tests - the walking tests (6-minute walk test and the incremental shuttle walking test) The step test will be performed on a 20 cm tall, single-step device with no handles. The criteria for stopping the test will be the same as described in standard operating procedures for the walking field tests, with the addition of the inability to follow the work rate for a period of 10 seconds.
  The main outcome of the test will be the highest number of steps and work rate achieved.

SUMMARY:
According to the official guidelines, a range of settings for cardiorespiratory rehabilitation, including the community- and home-based models, are considered to answer to the inadequate number of rehabilitation services, especially at hospitals, and, also, to respond to the patients' needs. For these settings outside the hospitals, new strategies for the assessment of exercise capacity and exercise training are essential. The modality of stepping can be a promising tool because it is inexpensive, portable, and reflects one of the main activities of daily living (stair climbing). The development of a new field test implies the establishment of normative values and reference equations generated from data of populations without disabilities to aim to characterize a defined population at a specific period of time, and evaluate and compare an individual's performance within a population.

DETAILED DESCRIPTION:
The primary aim of this project is to establish normative values and reference equations generated from Portuguese adults without disabilities of a new step test for the assessment of exercise capacity.

The investigators will perform a cross-sectional study in Portuguese adults (over 18 years) without disabilities. The study will be advertised at the university campus, surrounding areas, and interested participants can contact the research team for participation. The participants who agree will be seen by the principal investigator who will explain the nature of the study and assess eligibility for the study. The participants will sign informed consent.

For each participant, the study will be performed in one day. The participants will perform the incremental step test twice (30 minutes apart).

In addition, socio-demographic information (age and sex), anthropometric measures (weight, height, and body mass index), and clinical data (smoking status, comorbidities, and level of physical activity) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Portuguese nacionality
* Adults without disabilities aged >18 years
* Participants with body mass index between 18 and 30 kg/m2

Exclusion Criteria:

* Acute or chronic conditions (respiratory disease, cardiac disease, signs of cognitive or neuromuscular impairment, and significant musculoskeletal disorder)
* Conditions that could interfere with the ability to perform the step test
* Use of walking aids
* Post-symptomatic COVID-19 infected participants
* High-performance athletes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Portuguese adults (over 18 years) without disabilities will be included through an advertisement at the university campus and surrounding areas. Interested participants can contact the research team for participation. The participants who agree will be seen by the principal investigator who will explain the nature of the study and assess eligibility for the study. The participants will sign informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Number of steps | Through test completion, duration of the test 15 minutes
  The primary outcome will be the amount of steps performed in the step test

SECONDARY OUTCOMES:
Dyspnea during the tests | Through test completion, duration of the test 15 minutes
  Dyspnea experienced during the tests, monitored with the modified Borg scale, that ranges from 0 to 10, where 0 represents no dyspnea and 10 the worst dyspnea.
Fatigue during the tests | Through test completion, duration of the tests 15 minutes
  Fatigue experienced during the tests, monitored with the modified Borg scale, that ranges from 0 to 10, where 0 represents no fatigue and 10 the worst fatigue
Heart rate during the tests | Through test completion, duration of the tests 15 minutes
  Heart rate assessed during the tests, monitored with a cardiofrequencimeter
Oxygen saturation during the tests | Through test completion, duration of the tests 15 minutes
  Oxygen saturation assessed during the tests, monitored with a pulse oximeter

CONTACTS AND LOCATIONS:
Locations (1):
- Rui Vilarinho, Porto, Portugal